CLINICAL TRIAL: NCT02021747
Title: Biologic Basis Of Increased Susceptibility Of Smokers To Pulmonary Infection With Mycobacterium Tuberculosis
Status: Withdrawn | Type: Observational
Why Stopped: Research Changed Directions
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Other Study IDs: 14-00055 [JIRB]; NPRP 5-400-3-107 (Other: Qatar National Research Fund); 11262/11 (Other: HMC IRB)
Record Dates: First submitted 2013-11-22; First posted 2013-12-27 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Tuberculosis; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Tuberculosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Biological material from the lungs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Individuals with TB: Diagnosis of pulmonary tuberculosis without extra-pulmonary TB, confirmed by at least one of the following:
  1. Symptoms consistent with TB
  2. Chest X-rays and or chest CT consistent with TB
  3. Positive PPD test
  4. Positive sputum test
- Smokers: Active smoker as evidenced by self report and urine nicotine >30 ng/mL and urine cotinine >50 ng/mL
  Diagnosis of pulmonary tuberculosis without extra-pulmonary TB, confirmed by at least one of the following:
  1. Symptoms consistent with TB
  2. Chest X-rays and or chest CT consistent with TB
  3. Positive PPD test
  4. Positive sputum test
- Non-smokers: Never smokers is defined as someone who has smoked < 100 cigarettes per lifetime and whose urine nicotine <2 ng/mL and urine cotinine <5 ng/mL, at entry into the study
  Diagnosis of pulmonary tuberculosis without extra-pulmonary TB, confirmed by at least one of the following:
  1. Symptoms consistent with TB
  2. Chest X-rays and or chest CT consistent with TB
  3. Positive PPD test
  4. Positive sputum test
- Individuals with COPD: All study subjects should meet the "Lung Disease" protocol criteria for having COPD may be of any stage (GOLD I - IV), be ambulatory and have no evidence of respiratory failure
  Diagnosis of pulmonary tuberculosis without extra-pulmonary TB, confirmed by at least one of the following:
  1. Symptoms consistent with TB
  2. Chest X-rays and or chest CT consistent with TB
  3. Positive PPD test
  4. Positive sputum test

SUMMARY:
Identify a biologic (molecular) basis for the increased susceptibility of cigarette smokers to pulmonary TB (Mtb) by testing the hypothesis that smoking reprograms AM polarization towards a distinct phenotype associated with impaired host defense function against Mtb and that normalization of that phenotype via therapeutic modulation of the Alveolar Macrophage (AM) polarization or smoking cessation can restore the anti-Mtb host defense function of AM.

DETAILED DESCRIPTION:
Samples from Non-Smokers with TB, Smokers with TB and Smokers with COPD and TB will be collected in Qatar under JIRB 14-00055. All subjects will be undergoing a clinical bronchoscopy as part of their disease evaluation and will be asked to give additional samples for research. All "in vivo" processing of specimens from subjects with TB will be performed in Qatar. Mycobacterium tuberculosis infection (Mtb) continues to have a detrimental impact of public health worldwide. Based on the epidemiological evidence linking smoking, COPD and Mtb, and our preliminary data we hypothesize that smoking reprograms Alveolar Macrophages (AM) polarization towards a distinct phenotype associated with impaired host defense function against Myobacterium tuberculosis (Mtb) and that normalization of that phenotype via therapeutic modulation of the Alveolar Macrophages (AM) polarization or smoking cessation can restore the anti-Mtb host defense function of AM.

ELIGIBILITY:
Smokers and Non-smokers with TB

Inclusion Criteria:

* Must provide informed consent
* Current smokers and non-smokers
* Undergoing clinical bronchoscopy as required by their doctor for evaluation of their disease
* Diagnosis of pulmonary tuberculosis without extra-pulmonary TB, confirmed by at least one of the following:
* Symptoms consistent with TB
* Chest xray and or chest CT with TB
* Positive PPD test
* Positive sputum test

Exclusion Criteria:

* Females who are pregnant or nursing
* History of allergies to xylocaine, lidocaine, versed, valium, atropine, isoproterenol, terbutaline, aminophylline, or any local anesthetic

Smokers with TB and COPD

Inclusion Criteria:

* Must provide informed consent
* Current smokers with COPD
* Undergoing clinical bronchoscopy as required by their doctor for evaluation of their disease
* Diagnosis of pulmonary tuberculosis without extra-pulmonary TB, confirmed bu at least one of the following:
* Symptoms consistent with TB
* Chest xray and or chest CT consistent with TB
* Positive PPD test
* Positive sputum test

Exclusion Criteria:

* Non-smokers
* Females who are pregnant or nursing
* History of allergies to xylocaine, lidocaine, versed, valium, atropine, isoproterenol, terbutaline, aminophylline, or any local anesthetic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment will be from the referral base of the responsible investigator and other physicians, and review of admissions and hospital database. Patients, who may qualify for this study, will be identified by chart review, physician referral, and recruited by study investigators. The source of potential subjects will be the population of potential subjects with TB (smokers or non smokers), and with both TB and COPD, as defined before. Accrual will be random with no bias as to gender or racial/ethnic group.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Alveolar Macrophage | 1 week
  Changes in alveolar macrophage

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
All results of the proposed studies will be published in international peer-reviewed scientific journals, presented at meetings in Qatar, the regional and international conferences, and disseminated through the local Qatari media, seminars and lectures for high school and college students. The original data will be available to interested investigators using the conventional standards of biomedical science.